CLINICAL TRIAL: NCT00479570
Title: Phase 2A Multi-Centre, Double Blind, Placebo Controlled 3-Way Cross-Over Study To Investigate The Effect Of Single Doses Of PF-00446687 On Sexual Arousal And Sexual Desire In Women Suffering From Female Sexual Dysfunction (FSD).
Brief Title: Study To Investigate Effect Of A New Drug (PF-00446687) In Post-Menopausal Women Who Suffer From Sexual Dysfunction.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A8361015
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Female Sexual Dysfunction
MeSH Terms: interventions — 1-((1-tert-butyl-4-(2,4-difluorophenyl)pyrrolidin-3-yl)carbonyl)-3,5-dimethyl-4-phenylpiperidin-4-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study period 1, 2 or 3 (Experimental)
  Interventions: Drug: PF-00446687
- Placebo Study period 1, 2 or 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-00446687 — Single 200mg dose
  Arms: Study period 1, 2 or 3
Drug: Placebo
  Arms: Placebo Study period 1, 2 or 3

SUMMARY:
The purpose of this study is to investigate the effect of up to 200 mg of PF-00446687 on acute sexual arousal and sexual interest in post menopausal females, as well as examining the safety and toleration of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Women who have evidence of Female Sexual Arousal Disorder.
* Women who experience personal distress due to Female Sexual Dysfunction.
* Post menopausal women aged between 45 and 65 years.

Exclusion Criteria:

* Women whose sexual dysfunction is limited to certain types of stimulation, situation or specific partners.
* Women who experience pain with sexual intercourse or who have a sexual aversion disorder.
* Women suffering from female sexual dysfunction where the cause is treatable, for example inadequately controlled diabetes or thyroid dysfunction.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Assess effect of single doses of PF-00446687 on acute sexual arousal and sexual interest, using questionnaires, in post menopausal women suffering from Female Sexual Dysfunction. A diary will be completed for 7 days following the 3 dosing days. | From day of dosing until 7 days post-dose

SECONDARY OUTCOMES:
Assess effect of single doses on medium term (1 week) sexual arousal and interest. | Until 7 days post-dose
Assess variability of response and repeatability of design between 2 similar doses. | Comparison of response to be assessed until 7 days post dose
If possible assess the effect of PF-00446687 on vaginal blood flow on day 1 of each study period. | Day of dosing
Assess PK , safety and toleration on day 1 of each study period. | Day of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Kobenhavn OE, Denmark
- Pfizer Investigational Site, Oslo, Norway
- Pfizer Investigational Site, Danderyd, Sweden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8361015&StudyName=Study%20To%20Investigate%20Effect%20Of%20A%20New%20Drug%20%28PF-00446687%29%20In%20Post-Menopausal%20Women%20Who%20Suffer%20From%20Sexual%20Dysfunction.